CLINICAL TRIAL: NCT01279369
Title: The Use of Fetal Fibronectin (fFN) in Predicting Preterm Delivery Due to Abruptio Placenta in Patients With Minor Maternal Trauma.
Brief Title: The Use of Fetal Fibronectin to Predict Delivery Due to Abruptio Placenta
Status: Terminated | Type: Observational
Why Stopped: Quantitative assessment of fFN only able to be performed at one laboratory.
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, Wendy Kinzler, MD, Attending Physician, Winthrop University Hospital
Other Study IDs: 117104-4
Record Dates: First submitted 2011-01-14; First posted 2011-01-19 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Pregnancy Related; Trauma; Abruptio Placentae
Keywords: Pregnancy; Trauma; Placental Abruption; Fetal fibronectin
MeSH Terms: conditions — Wounds and Injuries; Abruptio Placentae

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fetal fibronectin
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine if the presence of fetal fibronectin in the cervicovaginal secretions of pregnant patients with minor maternal trauma predicts impending preterm delivery due to abruptio placenta.

DETAILED DESCRIPTION:
Optimal care of the pregnant trauma patient requires prompt and efficient care by a multidisciplinary team to evaluate both maternal and fetal status. Approximately 7% of pregnancies are complicated by trauma and traumatic injury remains the leading cause of non-obstetric maternal death.1-3 In the case of major or life-threatening trauma in pregnancy, assessment and stabilization of maternal cardiovascular and respiratory status is paramount and management is generally dictated by standard adult advanced cardiovascular support algorithms. In contrast, the evaluation and management of minor trauma in pregnancy is variable and often provider dependent.4-7 Regardless of the clinical and laboratory evaluation performed, the universal goal is to prevent maternal injury or death and optimize pregnancy outcomes.

Maternal trauma has been associated with adverse pregnancy outcome, including preterm labor, abruptio placenta, uterine rupture and fetal death.8, 9 Traditional trauma scoring systems correlate well with the severity of maternal injury and are useful in triaging the mother; however, these scoring systems have not been predictive of adverse pregnancy outcome.10,11 Major or life-threatening maternal trauma, which includes maternal shock, head injury resulting in coma, and emergency laparotomy for maternal indications is associated with a 40-50% fetal loss rate as compared to 1-5% in pregnant women after minor trauma. The risk of preterm labor after maternal trauma is increased 2-fold and the prevalence of abruptio placenta after minor blunt abdominal trauma is reported at 8%. 3,6-9,12

Upon initial evaluation in the obstetrical triage setting, the examination of maternal trauma patients is focused on detection of impending labor or abruptio placenta. This evaluation includes detailed history of the accident, physical examination, abdominal and transvaginal ultrasound to evaluate placental location and/or evidence of placental abruption and cervical length, external uterine contraction monitoring, continuous fetal heart rate monitoring and blood tests such as CBC, blood type, coagulation profile and Kleihauer-Betke staining. Although much has been written on the subject of trauma during pregnancy, there is little concrete data on objective measures which can be used to dictate triage and management decisions. A recent study by Cahill et al.13 has advocated for review of the extensive evaluations often performed after maternal trauma, specifically minor trauma, because they determined that none of the commonly used clinical and laboratory measures are predictive of adverse outcomes. Identification of laboratory measures predictive of impending delivery due to placental abruption will potentially enable physicians to individualize triage and evaluation of the maternal trauma patient, as well as direct treatment and management.

Fetal fibronectin is an extracellular matrix protein that is normally found in the fetal membranes and decidua.14 It is essentially an adhesive glycoprotein or "glue" at the maternal-fetal interface. In a normal pregnancy, fFN is undetectable in vaginal secretions from weeks 22 to 35. Disruption of the maternal-fetal interface causes the release of fFN into cervical and vaginal secretions. Detection of fFN before the normal onset of labor is an indicator of preterm birth risk, allowing opportunity to provide appropriate intervention. According to previous studies, the clinical utility of fFN lies in its negative predictive value. In non-trauma patients, the sensitivity of fFN in predicting impending delivery (within 7 days) is greater than 90%. A negative fFN result can be used to rule out impending deliver with greater than 99% certainty.15

Because abruptio placenta secondary to maternal trauma is the result of shearing forces separating the placenta from the uterine decidua, this outcome could potentially be predicted by a positive fFN result. This study is therefore undertaken to determine if the presence of fFN in cervicovaginal secretions is predictive of impending delivery or placental abruption in patients with maternal trauma. With better knowledge of the probable outcomes following maternal trauma and using the appropriate diagnostic and therapeutic modalities, optimal care following minor maternal trauma for the pregnant patient and fetus can be provided.

ELIGIBILITY:
Inclusion Criteria:

* Singleton intrauterine pregnancy ≥20 weeks and ≤35 weeks gestational age
* Chief complaint of minor maternal trauma including motor vehicle accident, patient fall or assault with absence of maternal conditions outlined in exclusion criteria

Exclusion Criteria:

* Maternal shock
* Unstable vital signs
* Altered sensorium
* Head injury resulting in coma
* signs or symptoms of intraperitoneal bleeding
* Emergency laparotomy for fetal or maternal indications
* Bone fractures
* History of previous abruptio placenta
* Known or suspected placenta previa
* Rupture of membranes
* Multiple gestation
* Advanced cervical dilatation ≥3cm
* Non-reassuring fetal status requiring intervention
* Vaginal bleeding on presentation
* History of intercourse and/or digital vaginal exam and/or vaginal ultrasound ≤24 hours prior to presentation
* Illicit drug use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for inclusion in the study are women aged 18 or over with singleton intrauterine pregnancy ≥20 weeks gestational age and ≤35 weeks gestational age presenting to the Winthrop University Hospital Labor & Delivery triage unit with a chief complaint of maternal trauma.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Delivery within 2 weeks of the trauma event | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wendy L. Kinzler, M.D., Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States